CLINICAL TRIAL: NCT03353064
Title: Telemedicine as a Proposed Solution Towards Efficiency of Healthcare Delivery for Einstein Pulmonary Patients on PAP/NIPPV for Hypercapnia
Brief Title: Telemedicine for Improving Outcome in Inner City Patient Population With Hypercapneic Respiratory Failure
Acronym: ETOUCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to recruit subjects
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Sunil Sharma, Division Chair and Program Director of Pulmonary, Critical Care, Allergy and Sleep Medicine, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ETOUCH Study
Record Dates: First submitted 2017-11-05; First posted 2017-11-27 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Hypercapnic Respiratory Failure; Chronic Obstructive Pulmonary Disease; Obesity Hypoventilation Syndrome; Sleep Disordered Breathing; Neuromuscular Diseases
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome; Sleep Apnea Syndromes; Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Statisticians will be receiving de-identified data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vivify + EMS (Active Comparator): This arm will have the Telemedicine kits and get scheduled EMS home visits. The subjects will complete daily biometrics / surveys / care plans through the telemedicine kit, as specified in the activity schedule Apart from the tablet device, EMS home visits will be scheduled on Day 7, Day 21 and Day 42 from discharge. During these home visits, the EM personnel will perform a check of the NIV/NIPPV device. They are able to adjust pressures according to your Pulmonologist / Sleep doctor's prescription, and troubleshoot any issues with the mask, the humidifier, etc. They will also measure End-tidal CO2 via nasal cannula.
  Interventions: Other: Vivify; Other: EMS
- Vivify Only (Active Comparator): This group will receive the telemedicine tablet and kit, with the same protocol as defined above.
  No EMS home visits will be set up
  Interventions: Other: Vivify

INTERVENTIONS:
Other: Vivify — A telemedicine kit will (Vivify) which will obtain daily biometrics (vital signs) and care plans. These are all monitored by the Pulmonary team remotely via an online portal. The telemedicine system has a set-up for alerts whenever there are clinical concerns (vital signs out of parameters), or non-use of the Non-invasive positive pressure ventilation (NIPPV). This system allows for video conferencing between the Pulmonary team (physician, respiratory therapist, nurse) to troubleshoot issues, and increase NIPPV compliance.
Other: EMS — Emergency medical service scheduled home visits for face to face troubleshooting of the NIPPV, environmental check and end-tidal CO2.
  Arms: Vivify + EMS

SUMMARY:
The Hypercapnia Telemedicine Outreach Program (E-TOUCH Study) aims to utilize telemedicine technology, as well as emergency medical services (EMS) home visits to address the problem with poor follow-up and compliance among Einstein's hypercapnic patients.

The hypothesis is that reaching out to the subjects' homes will allow more consistent healthcare delivery, increase healthcare efficiency and compliance with therapy, and overall decrease acute decompensated states / hypercapnic respiratory failure, decreasing ED visits and hospitalization.

DETAILED DESCRIPTION:
Hypercapnic respiratory failure is a prevalent medical problem, comprising a substantial number of ED visits and readmissions. The target population that are at high risk for developing hypercapnia are patients with obesity hypoventilation syndrome (OHS), chronic obstructive pulmonary disease (COPD), sleep disordered breathing (SDB) overlapping with COPD, and patients with neuromuscular disorders. These patients are commonly managed in the progressive care units or the intensive care unit for extended periods of time, which can over-utilize health systems resources. Einstein Medical Center's patient population includes multiple low-income communities / neighborhoods. Their educational background varies and constant education and counseling is an integral part of the treatment plan. These patients are particularly vulnerable due to a lack of geographic access and difficulty contacting healthcare providers via phone. Some of the patients may not be able to afford co-pays for clinic visits or are not able to follow up with a physician. In addition, patients treated with non-invasive ventilation in the hospital and require home therapy either never receive the device or are sub-optimally trained in its appropriate utilization. These patients may also be morbidly obese with mobility issues, which is another obstacle preventing patients from following up with their providers.

Positive airway pressure (PAP) therapy/ non-invasive positive pressure ventilation (NIPPV) are effective treatments to avoid acute hypercapnic respiratory failure; however, low compliance and poor follow-up are often recurring issues. These high-risk patients present in the emergency department acutely hypercapnic and encephalopathic with subsequent ICU admission and mechanical ventilation.This Telemedicine Outreach Program aims to utilize E-touch devices (Vivify-Go) in collaboration with home visits by EMS (Emergency medical services) to improve compliance and the efficiency of healthcare delivery. These efforts will hopefully lead to a decrease in acute decompensated respiratory states and hospital readmission rates.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years of age
* Evidence of hypercapnia (PCO2 ≥ 45mmHg) secondary to COPD-OSA overlap, OHS, Neuromuscular disease / weakness
* Requiring NIV / NIPPV outpatient
* Ability to operate a smart device / tablet
* Informed consent

Exclusion Criteria:

* Non-English or Non-Spanish- speaking (device videos and surveys are available in English or Spanish only)
* Patients unable to give consent
* Pregnant women
* Prisoners
* Patients <18 years of age
* Patient already on NIPPV/ CPAP at home and compliant on therapy
* Significant non-pulmonary conditions (CHF with EF < 40%), Pulmonary hypertension with PASP> 60 mmGH, severe valvular heart disease, end-stage renal disease or end-stage liver disease.
* Patients without health insurance
* Residing out of state (Pennsylvania)
* Patients with current or history of drug / narcotic dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
30-day ED and Hospital readmission Rate | 30 days
  Patients are followed from enrollment for the next 30 days. We will compare rate of re-admissions between the 2 parallel intervention arms, and check the p-value

SECONDARY OUTCOMES:
SF-12 questionnaire | every 2 weeks for duration of 6 weeks
  The SF-12 questionnaire gives an assessment score of subject's mental and physician functioning and overall health-related quality of life. We will compare scores of subjects in the parallel intervention groups
NIV compliance | 6 weeks
  This is a YES or NO determination of NIV compliance using the CMS (Centers of Medicare and Medicaid) criteria of at least 4hrs use of NIV per day, at least 70% of a 30-day period. We will compare the number of compliant against non-compliant subjects in the 2 parallel intervention groups

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, Principal Investigator — Albert Einstein Medical Center
Locations (1):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Cruz,Rebecca, Harman Saman, Olliver O'Sullivan, Norashikin Amran, Jumaa Bwika, Ben Beauchamp, Rahul Mukherjee. "Readmission and mortality after first hospital admission with acute hypercapnic respiratory failure (AHRF) requiring non-invasive ventilation (NIV)" European Respiratory Journal (2013) 42:P2490
- [Background] Konikkara J, Tavella R, Willes L, Kavuru M, Sharma S. Early recognition of obstructive sleep apnea in patients hospitalized with COPD exacerbation is associated with reduced readmission. Hosp Pract (1995). 2016;44(1):41-7. doi: 10.1080/21548331.2016.1134268. Epub 2016 Jan 20. PMID 26691510
- [Background] Riachy M, Najem S, Iskandar M, Choucair J, Ibrahim I, Juvelikian G. Factors predicting CPAP adherence in obstructive sleep apnea syndrome. Sleep Breath. 2017 May;21(2):295-302. doi: 10.1007/s11325-016-1408-y. Epub 2016 Sep 16. PMID 27638725
- [Background] Taylor Y, Eliasson A, Andrada T, Kristo D, Howard R. The role of telemedicine in CPAP compliance for patients with obstructive sleep apnea syndrome. Sleep Breath. 2006 Sep;10(3):132-8. doi: 10.1007/s11325-006-0059-9. PMID 16565867
- [Background] Turino C, de Batlle J, Woehrle H, Mayoral A, Castro-Grattoni AL, Gomez S, Dalmases M, Sanchez-de-la-Torre M, Barbe F. Management of continuous positive airway pressure treatment compliance using telemonitoring in obstructive sleep apnoea. Eur Respir J. 2017 Feb 8;49(2):1601128. doi: 10.1183/13993003.01128-2016. Print 2017 Feb. PMID 28179438
- [Result] Bruyneel M. Technical Developments and Clinical Use of Telemedicine in Sleep Medicine. J Clin Med. 2016 Dec 13;5(12):116. doi: 10.3390/jcm5120116. PMID 27983582